CLINICAL TRIAL: NCT06129084
Title: ctDNA-FGFR Status as a Predictive Biomarker for FGFR Targeted Therapy
Brief Title: A Study to Compare the Results of FGFR Testing by Either ctDNA Blood Testing or Standard Tumor Tissue Testing
Status: Active, not recruiting | Type: Observational
Sponsor: Bernie Eigl (Other)
Collaborators: Vancouver Prostate Centre (Other); Lady Davis Institute (Other); Bladder Cancer Canada (Unknown)
Responsible Party: Sponsor-Investigator, Bernie Eigl, Principal Investigator, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Other Study IDs: ctDNA FGFR
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Bladder Cancer; Metastatic Urothelial Carcinoma
Keywords: ctDNA-FGFR; FGFR Biomarker; Erdafitinib
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma ctDNA and archival tumour tissue will be tested for FGFR status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Bladder Cancer: Patients with metastatic bladder cancer who will have archival tissue sent for FGFR testing.
  Interventions: Genetic: FGFR Testing

INTERVENTIONS:
Genetic: FGFR Testing — Determine whether ctDNA testing for FGFR provides the same results as the standard tissue testing.

SUMMARY:
A new drug, erdafitinib, became available for some patients with bladder cancer that has spread to other organs. To qualify, patients must have specific genetic changes in their tumors. Currently, doctors use tumor tissue samples to check for these genetic changes, but these samples might not accurately reflect the current state of the patient's cancer.

In this study, Investigators will test the patient's blood for these genetic changes in addition to the tumor tissue samples. It is thought that the blood test will give a more accurate result.

Investigators hope this study will help to find out if more patients can benefit from erdafitinib than the ones identified by tissue testing only.

DETAILED DESCRIPTION:
Recently, the first targeted therapy for patients with metastatic urothelial cancer (mUC) received approval, i.e. erdafitinib. Erdafitinib is a pan-FGFR small molecule inhibitor. Approximately twenty percent of mUC patients' tumors harbor qualifying alterations in FGFR2 or FGFR3. Currently, standard testing uses archival tumor tissue. However, this type of testing may not be representative of a patient's clinically dominant tumor clone at the time of treatment initiation due to temporal and spatial biopsy bias of archival tissue testing.

In this study, patients will undergo circulating tumor DNA testing, in addition to conventional tissue testing, for treatment eligibility. Investigators hypothesize that blood-based ctDNA testing will provide a more accurate assessment of somatic FGFR status than same patient archival primary tissue.

This study's objectives are:

Objective 1 (Primary): To evaluate the diagnostic value of ctDNA testing against the "gold standard" of tissue testing.

Objective 2 (Secondary): To evaluate whether ctDNA may be a superior predictive marker by identifying actionable FGFR alterations that are currently missed on tissue assays.

Procedures:

* Medical history will be reviewed, including all previous anti-cancer treatments.
* A blood sample will be collected for ctDNA testing at the time of screening for FGFR alterations and at progression under erdafitinib therapy. Test results will be compared to archival tissue testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic bladder cancer who are about to undergo tissue testing for FGFR mutations and who have blood samples drawn during the management of their disease are eligible to be included in this analysis.

Exclusion Criteria:

* Metastatic bladder cancer patients who will not have tissue sent for FGFR testing will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic urothelial cancer who are screened for erdafitinib eligibility as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic value of ctDNA testing against standard tissue testing | For the primary objective, a single blood sample is collected at the time of screening for treatment eligibility
  Investigators will evaluate ctDNA as a diagnostic test against the de facto gold standard of tissue testing.

SECONDARY OUTCOMES:
To evaluate whether ctDNA may be a superior predictive marker by identifying actionable FGFR mutations that are currently missed on tissue assays | For this secondary objective, a single blood sample is collected at the time of screening for treatment eligibility
  To quantify the additional value of ctDNA testing, Investigators will calculate the percentage of eligible patients based on ctDNA testing among conventional testing ineligible or "negative" patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Eigl, Study Chair — British Columbia Cancer Agency; Alexander Wyatt, Study Chair — Vancouver Prostate Centre
Locations (7):
- Canada (7):
  - Arthur J.E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHU de Québec-Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
No plans for future use of the data at this point. Only the study Principal Investigator will have access to the data in the future.

REFERENCES:
- [Background] Knowles MA, Hurst CD. Molecular biology of bladder cancer: new insights into pathogenesis and clinical diversity. Nat Rev Cancer. 2015 Jan;15(1):25-41. doi: 10.1038/nrc3817. PMID 25533674
- [Background] Loriot Y, Necchi A, Park SH, Garcia-Donas J, Huddart R, Burgess E, Fleming M, Rezazadeh A, Mellado B, Varlamov S, Joshi M, Duran I, Tagawa ST, Zakharia Y, Zhong B, Stuyckens K, Santiago-Walker A, De Porre P, O'Hagan A, Avadhani A, Siefker-Radtke AO; BLC2001 Study Group. Erdafitinib in Locally Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2019 Jul 25;381(4):338-348. doi: 10.1056/NEJMoa1817323. PMID 31340094